CLINICAL TRIAL: NCT01921426
Title: A Phase 1 Dose Escalation Study of GC4419 in Combination With Radiation and Chemotherapy for Squamous Cell Cancers of the Head and Neck.
Brief Title: A Phase 1 Dose Escalation Study of GC4419 in Combination With Chemoradiation for Squamous Cell Cancer of the Head & Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GT-001
Record Dates: First submitted 2013-08-08; First posted 2013-08-13 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity; Squamous Cell Carcinoma of the Oropharynx
Keywords: Squamous Cell Carcinoma of the Head and Neck; Oral Cavity; Oropharynx; Radiation; Chemotherapy; Cisplatin; Oral Mucositis; Superoxide Dismutase
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Stomatitis | interventions — avasopasem manganese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GC4419 (Experimental): Open label, dose escalation study of GC4419 administered in 14 doses, corresponding to the first 14 doses of radiation therapy. Each dose will be given intravenously over 60 minutes. The possible doses which may be tested are: 15mg, 30mg, 50mg, 75mg, 112mg, and 170mg.
  Interventions: Drug: GC4419

INTERVENTIONS:
Drug: GC4419 — GC4419 is a novel, highly stable manganese-containing macrocyclic ligand complex with a molecular weight of 483, whose activity mimics that of naturally occurring superoxide dismutase (SOD) enzymes. It is therefore a prototype of a new class of drugs termed selective SOD mimetics. GC4419 selectively removes superoxide anions without reacting with other reactive oxygen species, including nitric oxide, hydrogen peroxide, and peroxynitrite.

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and the highest dose of GC4419 that can be given to patients with squamous cell cancer of the head and neck who are receiving standard radiation therapy and chemotherapy. This study will also evaluate GC4419 for the following:

* Effect on the incidence and severity of radiation induced oral mucositis;
* Effect on the response rate of squamous cell cancer of the head and neck who are receiving radiation therapy and chemotherapy;
* Total concentrations of GC4419 that can be achieved in the blood;
* Changes in proteins and genetics associated with oral mucositis;
* Impact on delayed toxicities of radiation (dry mouth and reduced ability to fully open the mouth);
* Observe changes in genetic and molecular markers of oral mucositis;
* Observe the usage of extra health resources (e.g., unplanned ER visits, feeding tube use, etc.) of study patients;
* Assess the overall quality of life in study patients with oral mucositis.

DETAILED DESCRIPTION:
This is a multi-center, single-agent, open-label clinical trial to be conducted in serial cohorts of patients with squamous cell cancer of the head and neck receiving escalating doses of GC4419 in combination with standard chemoradiation.

The study will follow a standard 3+3 cohort design typical for phase I clinical trials, in which 3 patients are initially entered at a given dose level and observed for dose-limiting toxicity (DLT). For the purposes of managing dose escalation, the DLT observation window will be defined as the first dose of GC4419 through 24 hours following the last dose of GC4419 for an individual patient. If zero of three patients in a dose cohort experience a DLT during the DLT observation window, enrollment to the next higher dose level will begin. If 1 of 3 patients experiences a DLT within the DLT observation window, 3 additional patients will be added to the dose level. If no DLTs are observed in the 3 additional patients, dose escalations will resume with enrollment to the next higher dose level. If ≥2 patients in a cohort experience a DLT within the DLT observation window, that dose will be considered to have exceeded the MTD. The MTD is defined as the highest dose where ≤ 1 of 6 patients experience a DLT during the DLT observation period.

Decisions to expand a dose cohort or proceed to dose escalation will be made after review of the safety data at a dose level by the Sponsor in collaboration with investigators and appropriately qualified consultants, as needed.

Planned dose levels will be 15, 30, 50, 75, 112, 150, 175, 210, and 250 mg/day, with subsequent dose increments of 50 mg/day, as data warrant or until an MTD is determined. These dose levels represent maximum dose escalation increments. At any time, if ongoing review of safety and other data warrant, intermediate dose levels may be studied (with 3-6 patients enrolled per dose level). These intermediate dose levels may be selected below the next planned dose level or between two dose levels previously studied. If an MTD has not been determined after the 250 mg dose level, further dose escalation may be undertaken at increments of 50 mg/day.

Initial dose escalation will proceed on a treatment schedule wherein GC4419 is administered prior to IMRT on each of the first 14 scheduled days of IMRT. Separate dose cohorts will also be studied wherein GC4419 is administered on each of the first 20, 25, 30, or all 35 days of IMRT (four, five, six, or seven weeks of Active Treatment). Daily dosing of GC4419 by this schedule will begin at a dose that has been shown not to exceed the MTD by the original, 14-dose schedule. Further dose levels may be selected following the same planned dose level guidelines (including possible intermediate dose levels) and rules for determining an MTD as for the 14-dose schedule. At a given daily dose level, extension of the dosing period may be undertaken in increments of one week (5 doses, M-F) per cohort, in successive cohorts. For example, dosing for 20 doses (4 weeks) may proceed at a given dose level only if the MTD has not been exceeded for the same daily dose given for 14 doses; or, dosing for 25 doses (5 weeks) may proceed at a given daily dose level only if the MTD has not been exceeded for the same daily dose given for 20 doses (4 weeks); etc. Note again that, for any cohort and treatment duration, the DLT observation period will extend to 24 hours after the last GC4419 dose for an individual patient. Note also that an extension of dosing duration and an escalation of the daily dose in the same step is not permitted.

In addition, a separate dosing cohort may be concurrently enrolled to receive 30 mg/day, M-F, for 35 doses (7 weeks), based on the calculation that the total dose administered to a given patient (1050 mg) will not exceed the total dose received by 3 patients at 75 mg/d x 14 doses (1050 mg), which was previously determined to be safe (i.e., without any patients having experienced a DLT). If this dose and schedule does not exceed the MTD as defined in this protocol, enrollment of additional 7-week dosing cohorts may be undertaken by applying the same total dose approach to future dose levels administered for <7 weeks without exceeding the MTD.

On the 14-day schedule, missed doses of GC4419 may be made up prior to study day 28. On schedules employing administration of GC4419 for 20 or more doses, M-F, no GC4419 doses will be made up.

On any schedule, additional patients may be studied at dose levels not exceeding the MTD to characterize the safety, pharmacokinetics, and potential efficacy of GC4419 at those dose levels.

At least one recommended Phase 2 dose, by at least one schedule, will be identified for GC4419. More than one dose may be identified for further assessment of exposure/response relationships. Dose(s) recommended for further study will be at or below the MTD, with exposure and preliminary efficacy data suggesting that they may warrant further investigation for safety and efficacy.

Treatment will be administered on an outpatient basis. Supportive care measures including those directed at controlling symptoms resulting from the patient's malignancy are allowed at the discretion of the treating investigator.

Pharmacokinetic samples will be obtained from all patients.

Primary Objectives:

1. To assess the safety and tolerability of GC4419 when administered with standard chemoradiation, by observation of the frequency and severity of adverse events with the study regimen
2. To determine a Maximum Tolerated Dose/Recommended Phase 2 dose and schedule of GC4419 for further study when administered in combination with standard chemoradiation to patients with squamous cell cancers of the mouth and oropharynx

Secondary Objectives:

1. To determine the pharmacokinetic profile of GC4419 when administered in combination with standard chemoradiation
2. To determine the incidence, severity, time to first onset and duration of oral mucositis in patients receiving GC4419 when administered in combination with standard chemoradiation
3. To preliminarily assess the tumor response to standard chemoradiation when administered in conjunction with GC4419

Exploratory Objectives:

1. To determine the pharmacodynamic effects of GC4419
2. To correlate pharmacokinetic and pharmacodynamic effects of GC4419 with the incidence, severity and time to first onset of oral mucositis
3. To evaluate the potential synergistic effect of GC4419 with chemoradiation on tumor response using pharmacokinetic and pharmacodynamic analyses
4. To evaluate the effect of GC4419 on specific late toxicities (xerostomia and trismus) of standard chemoradiation
5. To collect information about health resource utilization
6. To collect information about health-related quality of life (Oral Mucositis Daily Questionnaire)

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-confirmed diagnosis of squamous cell carcinoma of the head and neck (SCCHN), defined as SCC of the oral cavity or oropharynx, that will be treated with standard cisplatin and Intensity-Modulated Radiation Therapy (IMRT)
* Males or females aged 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate bone marrow, liver and kidney function
* Negative serum pregnancy test for females of childbearing potential
* Properly obtained written informed consent

Exclusion Criteria:

* Tumor of the lips, larynx, hypopharynx, nasopharynx, sinuses, salivary glands or unknown primary tumor
* Metastatic disease (Stage IV C)
* Prior chemotherapy for SCCHN and/or radiotherapy to the region of the study cancer or
* Receiving any agent classified as an antioxidant
* History of malignant tumors other than SCCHN within the last 5 years, except non-melanoma skin cancer or curatively excised in situ cervical carcinoma
* Active infectious disease excluding oral candidiasis
* Presence of oral mucositis at study entry
* Chronic immunosuppression
* Known history of HIV or active hepatitis B/C )
* Prior history of hearing impairment
* Use of investigational agent within 30 days of study entry
* Known allergies or intolerance to cisplatin and similar platinum-containing compounds
* Requirement for concurrent treatment with nitrates or other drugs that may, in the judgment of the treating investigator, create a risk for a precipitous decrease in blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Frequency and Severity of Adverse Events Resulting from GC4419 | 14 - 35 days
  GC4419 will be evaluated to determine safety, tolerability, and the maximum tolerated dose of GC4419 that can be administered to patients with squamous cell cancer of the head and neck who are receiving concurrent radiation (50-70 Gy, administered daily x 5 [M-F], in 2.0-2.2 Gy fractions) and chemotherapy (cisplatin, 80-100mg/m2, q3 weeks or weekly cisplatin 30-40mg/m2 x 6 weeks). Patients will receive 14 - 35 doses of GC4419 in serially ascending cohorts for dose and duration, which correspond to the first doses of radiation, schedule dependent. Dose limiting toxicity will be evaluated through 24 hours following the last dose of GC4419.

SECONDARY OUTCOMES:
Rate and Extent of Exposure to GC4419 (Pharmacokinetic Profile) | 18 - 49 Days
  Determine the pharmacokinetic profile, including the extent and rate of exposure (e.g., maximum concentration, total exposure, half life, time to maximum concentration, accumulation, etc.) to GC4419, as well as GC4419 kinetics (e.g., half-life, in patients with squamous cell carcinoma of the head and neck receiving GC4419 when administered in combination with standard chemoradiation.
Oral Mucositis | 49 Days
  Determine the incidence, severity, time to first onset and duration of oral mucositis in patients with squamous cell carcinoma of the head and neck receiving GC4419 when administered in combination with standard chemoradiation.
Antitumor Effect | 14 Months
  Preliminarily assess the tumor response to standard chemoradiation when administered in conjunction with GC4419 at approximately 1 year following completion of chemoradiation.

OTHER OUTCOMES:
Pharmacodynamic Profile | 49 Days
  Determine the pharmacodynamic profile of GC4419 in patients with squamous cell carcinoma of the head and neck receiving GC4419 when administered in combination with standard chemoradiation by observing the changes in proteins and genetic markers associated oral mucositis.

CONTACTS AND LOCATIONS:
Overall Officials: Jon T. Holmlund, MD, Study Director — Galera Therapeutics, Inc.; Madhavi Venigalla, MD, Principal Investigator — Lakeland Regional Cancer Center; Weining Zhen, MD, Principal Investigator — University of Nebraska; Douglas Adkins, MD, Principal Investigator — Washington University School of Medicine; Pardip Pathare, MD, Principal Investigator — Norwalk Hospital; Sanjiv Agarwala, MD, Principal Investigator — St. Luke's Cancer Center; Charles Kunos, MD, PhD, Principal Investigator — Summa Health System- Cooper Cancer Center; Yuhchyau Chen, MD, PhD, Principal Investigator — University of Rochester; John Buatti, MD, Principal Investigator — University of Iowa; Aftab Mahmood, MD, Principal Investigator — Cancer Specialists of South Texas, P.A.; Larisa Greenberg, MD, Principal Investigator — West Penn Allegheny Health System; Marcelo Bonomi, MD, Principal Investigator — Wake Forest University Health Sciences; Christopher M Lee, MD, Principal Investigator — Cancer Care Northwest
Locations (10):
- United States (10):
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - University of Iowa, Iowa City, Iowa
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Rochester Medical Center, Rochester, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Summa Health System- Cooper Cancer Center, Akron, Ohio
  - St. Luke's Cancer Center, Easton, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Cancer Care Northwest, Spokane, Washington